CLINICAL TRIAL: NCT00308776
Title: Effect of Cholecystokinin on Binge Eating in Bulimia Nervosa
Brief Title: Cholecystokinin for Reducing Binge Eating in People With Bulimia Nervosa
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit subjects
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: #4736; DATR A2-AID
Record Dates: First submitted 2006-03-28; First posted 2006-03-30 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2012-05

CONDITIONS: Bulimia Nervosa; Eating Disorders
MeSH Terms: conditions — Bulimia Nervosa; Feeding and Eating Disorders | interventions — Cholecystokinin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cholecystokinin (Experimental): Participants will receive intravenous saline plus cholescystokinin.
  Interventions: Procedure: Cholecystokinin (CCK) infusion
- Saline (Placebo Comparator): Participants will receive intravenous saline only.
  Interventions: Procedure: Saline infusion

INTERVENTIONS:
Procedure: Cholecystokinin (CCK) infusion — Participants will begin infusion with a normal saline solution. After 10 minutes of saline infusion, participants will eat a small bowl of tomato soup, followed 20 minutes later by a 15-minute infusion of saline plus CCK.
  Arms: Cholecystokinin
Procedure: Saline infusion — Participants will begin infusion with a normal saline solution. After 10 minutes of saline infusion, participants will eat a small bowl of tomato soup, followed 20 minutes later by a 15-minute infusion of saline only.
  Arms: Saline

SUMMARY:
This study will determine the effectiveness of administrating a dose of cholecystokinin during a binge eating episode in reducing this eating behavior in people with bulimia nervosa.

DETAILED DESCRIPTION:
Bulimia Nervosa (BN) is a serious eating disorder that is characterized by frequent uncontrolled eating binges. These binges are often followed by compensatory behavior, including the following: self-induced vomiting; misuse of laxatives, diuretics, enemas, or other medications to induce purging; fasting; or excessive exercise. If left untreated, BN can lead to many serious health issues: tooth decay; irregular menstruation; bowel damage; constipation; heart and kidney disease; intestinal damage; puffiness, especially in the face and fingers; increased hair growth on the face and body; and mineral imbalances in the body. Cholecystokinin (CCK) is a hormone that is released by the small intestine, and functions as a trigger for digestion and hunger suppression. People with BN often have disturbances in the release of CCK, which may contribute to their binge eating behavior. This study will determine the effectiveness of administrating a dose of CCK during a binge eating episode in reducing this eating behavior in people with BN.

This study will enroll females with BN and healthy females without BN. Interested participants will first report to the study site for an interview about their feelings on their eating habits. If eligible, participants will report to the study site at 9 A.M. on 4 days. Upon arrival, they will receive a standardized breakfast of apple juice and an English muffin with butter. Participants will then return 2.5 hours later to start an IV and begin infusion with a normal saline solution. After 10 minutes of saline infusion, participants will eat a small bowl of tomato soup, followed 20 minutes later by a 15-minute infusion of either saline or saline plus CCK. Participants will then be given a meal of macaroni and beef. They will be alone in the room while eating, but will be monitored by TV camera. Nothing, however, will be taped or recorded. A tape recording will be used to instruct participants when to begin eating. Participants will be instructed to either eat until an assistant returns to the room, or eat as much as they can. Participants will also fill out questionnaires before and after each meal, and sometimes during a meal. The amount of food consumed after an infusion with CCK will be assessed upon study completion.

For information on related studies, please follow these links:

http://clinicaltrials.gov/show/NCT00307190

http://clinicaltrials.gov/show/NCT00304187

ELIGIBILITY:
Inclusion Criteria for Patients with BN:

* Meets DSM-IV criteria for BN
* BN duration of more than 1 year
* Self-induces vomiting
* Weighs between 80 and 120% of ideal body weight

Exclusion Criteria for Patients with BN:

* Significant medical illness
* Current or lifetime history of schizophrenia, bipolar disorder, or other psychotic disorder, as defined by DSM-IV-TR criteria
* Current DSM-IV-TR diagnosis of organic mental disorder, factitious disorder, or malingering
* History of a personality disorder (e.g., schizotypal, borderline, or antisocial) that might interfere with the study procedures
* At risk for suicide, as defined by the expression of an imminent plan or attempt within the 6 months prior to study entry
* Currently taking psychotropic medications or medications that affect gastrointestinal function
* Moderate to severe depression, as defined by a score of greater than 28 on the Hamilton Depression Rating Scale
* Drug or alcohol abuse within the 3 months prior to study entry
* Pregnant, planning to become pregnant, or lactating
* Body mass index (BMI) of less than 18 (underweight)

Inclusion Criteria for Normal Weight Controls:

* No current or past psychiatric history
* No history of binge eating or vomiting
* 80-120% of ideal body weight

Exclusion Criteria for Normal Weight Controls:

* Significant medical illness
* Current psychotropic medications and current medications that affect GI function
* Drug or alcohol abuse in last 3 months
* Pregnancy, planning to become pregnant or laction

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2003-10; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Amount of food consumed after administration of CCK (measured upon study completion) | Measured at Day 4

CONTACTS AND LOCATIONS:
Overall Officials: B. Timothy Walsh, MD, Principal Investigator — New York State Psychiatric Institute at Columbia University Medical Center
Locations (1):
- New York State Psychiatric Institute, New York, New York, United States